CLINICAL TRIAL: NCT06954766
Title: A Randomized, Double-blind, Sham-controlled, Initial Pilot Study to Evaluate the Safety and Temporary Symptom Improvement Efficacy of CKD-981 in Patients With Degenerative Knee Osteoarthritis
Brief Title: Initial Pilot Study to Evaluate the Safety and Temporary Symptom Improvement Efficacy of CKD-981
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A145_01OA2401
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Knee Osteoarthritis
Keywords: CKD-981
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Expermental group 1 (Experimental): Patients assigned to this group will receive treatment with the medical device CKD-981(1) in combination with a placebo.
  Interventions: Device: CKD-981(1); Drug: Placebo Drug
- Expermental group 2 (Experimental): Patients assigned to this group will receive treatment with the medical device CKD-981(2) in combination with a placebo.
  Interventions: Device: CKD-981(2); Drug: Placebo Drug
- Sham group (Sham Comparator): Patients assigned to this group will receive treatment with the sham device in combination with a placebo.
  Interventions: Device: Sham device; Drug: Placebo Drug
- Reference group (Sham Comparator): Patients assigned to this group will receive treatment with the sham device in combination with a reference drug.
  Interventions: Device: Sham device; Drug: Reference Drug

INTERVENTIONS:
Device: CKD-981(1) — 20 minutes per day, 5 days a week for 6 weeks.
  Other Names: Expermental Device 1
  Arms: Expermental group 1
Device: CKD-981(2) — 20 minutes per day, 5 days a week for 6 weeks.
  Other Names: Expermental Device 2
  Arms: Expermental group 2
Device: Sham device — 20 minutes per day, 5 days a week for 6 weeks.
  Other Names: CKD-981 Sham Device
  Arms: Reference group; Sham group
Drug: Reference Drug — QD for 6 weeks
  Other Names: NSAIDs
  Arms: Reference group
Drug: Placebo Drug — QD for 6 weeks
  Other Names: Placebo for NSAIDs
  Arms: Expermental group 1; Expermental group 2; Sham group

SUMMARY:
The purpose of this study is to prove that the temporary symptom improvement effect on knee osteoarthritis using CKD-981

DETAILED DESCRIPTION:
The aim of this pilot study is to evaluate the efficacy and safety of CKD-981 in patients with mild to moderate degenerative knee osteoarthritis who have been experiencing pain more than 8 weeks

ELIGIBILITY:
Inclusion Criteria:

* Patients between 40 years and 80 years old
* Patients who have experiencing knee pain more than 8 weeks
* VAS more than 40 mm
* Kellgren and Lawrence grade 2 and 3 in X' ray knee joint

Exclusion Criteria:

* Previous knee surgery in affected side
* Patients with Rheumatoid arthritis, connective tissue disease, Paget's disease
* Infection of knee joint
* BMI more than 35kg/m2

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-12 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change in weight-bearing knee pain measured using the Visual Analog Scale(VAS) | 6 Weeks
  Pain will be measured using a 10-cm Visual Analog Scale (VAS), with scores ranging from 0 (no pain) to 10 (worst imaginable pain)

SECONDARY OUTCOMES:
Change in weight-bearing knee pain measured using the Visual Analog Scale(VAS) | 2 weeks, 4 weeks
  Pain will be measured using a 10-cm Visual Analog Scale (VAS), with scores ranging from 0 (no pain) to 10 (worst imaginable pain)
Change in total K-WOMAC (Korean Western Ontario and McMaster Universities Osteoarthritis Index) score from baseline | 2 weeks, 4 weeks, 6 weeks
  The K-WOMAC consists of 24 items, with each item scored on a 5-point scale (0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe), where higher scores indicate greater symptom severity

CONTACTS AND LOCATIONS:
Locations (1):
- Wonju Severance Christian Hospital, Wŏnju, South Korea

IPD SHARING:
Plan to Share IPD: No